CLINICAL TRIAL: NCT02077985
Title: Sensory Adapted Dental Environment to Enhance Oral Care for Children With Autism
Brief Title: Sensory Adapted Dental Environment to Enhance Oral Care for Children With ASD
Acronym: SADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Sharon Cermak, Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5R34DE022263-02 (NIH)
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Autism
Keywords: autism; electrodermal activity; cooperation; anxiety; distress; stress; oral care; sensory processing; behavior; occupational therapy
MeSH Terms: conditions — Autistic Disorder; Anxiety Disorders; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Dental Environment (No Intervention): There are two dental environments - the regular dental environment and the sensory dental environment; each child will be randomized to which is first. In the Regular dental environment no sensory characteristics of the dental environment are altered, the cleaning is conducted as per usual.
- Sensory Adapted Dental Environment (Experimental): There are two dental environments - the regular dental environment and the sensory dental environment; each child will be randomized to which is first. In the Sensory Adapted Dental Environment the sensory characteristics of the dental environment are altered (visual, auditory, tactile adaptations).
  Interventions: Behavioral: Sensory Adapted Dental Environment

INTERVENTIONS:
Behavioral: Sensory Adapted Dental Environment — See study arm description.
  Arms: Sensory Adapted Dental Environment

SUMMARY:
The goal of this project is to collect information that will support a later clinical trial on the effectiveness of a specially adapted dental environment for children who have difficulty tolerating oral care in the dental clinic. We hypothesize that adapting the sensory environment in the dental office by modifying the sounds, sights, smells and tactile experiences will result in decreased anxiety, increased cooperation, and fewer behavior problems for children with Autism Spectrum Disorders, and to a lesser extent for typically developing children especially those who have dental anxieties. This has the potential contribute to increased child comfort as well as safer, more efficient, and less costly treatment for a large population, as potentially more than one-fourth of all children may benefit from a sensory adapted dental environment.

DETAILED DESCRIPTION:
The goal of this R34 NIDCR Planning and Pilot Data Grant is to collect information to support a later clinical trial on the effectiveness of a specially adapted dental environment for children who have difficulty tolerating oral care in the dental clinic. Within this project, two groups of children were studied: children with autism spectrum disorders (ASD) and typically developing children, including those who are over-reactive to sensory stimulation. Commonly, such children exhibit anxiety and negative behavioral reactions when confronted with experiential aspects of dental visits such as exposure to bright fluorescent lighting, touch in or around the mouth, or the texture and smell of various oral care products. We pilot tested a sensory adapted dental environment (SADE) to examine its effect on reducing anxiety and behavioral problems among the targeted groups of children. The SADE intervention includes such adaptations as dimmed lighting, exposure to soothing music, and application of a special vest which provides deep pressure sensations that are calming. If our preliminary assessment produces promising results, we will later more comprehensively test the intervention in a full-scale randomized clinical trial, which will be supported by a U01 award.

The specific aims of the R34 grant are to promote the ability to conduct the future trial by:

1. Developing a manual for the SADE intervention and assessing the intervention's feasibility.
2. Collecting preliminary data on the intervention's effectiveness and potential cost-savings.
3. Pilot testing the recruitment strategy and assessment battery that will be used in the anticipated trial.
4. Developing the system of documents and data management for the future trial.
5. Generating the proposal for the U01 award to conduct the planned trial.

Research participants were 45 ethnically diverse children aged 6-12 years, 22 with ASD and 23 who are typically developing. Each child underwent two dental cleanings four months apart: dental cleaning in a standard dental environment and dental cleaning in the sensory adapted environment. For each group of children (i.e., ASD and typically developing), these two conditions were compared in their effects on anxiety and negative behavioral reactions, as measured by videotape coding, psychophysiological indices, and various rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism using ADOS (or) typically developing
* age 6 to 12
* parents speak English or Spanish
* in need of an oral cleaning (no previous cleaning within past four months)

Exclusion Criteria:

* disability such as cleft palate, significant motor impairment (e.g cerebral palsy), no genetic, endocrine, or metabolic dysfunction that would interfere with oral care or EDA.

Additional exclusion for participants in Typical Group include

* diagnosis of ASD or other DD
* diagnosis of ADHD, anxiety disorder, bipolar disorder
* siblings not diagnosed with ASD

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Electrodermal activity (EDA) | Recorded continuously for three minutes prior to cleaning, through duration of cleaning (approximately 10-45 minutes), and for three minutes at end of cleaning for each dental cleaning.
  Electrodermal activity (EDA) is a non-invasive measure of the ability of the skin to conduct an electrical current, which increases when the sympathetic "fight or flight" nervous system is activated during times of stress. EDA was analyzed in two ways in this study to investigate physiological stress/anxiety: (1) tonic skin conductance level (SCL) and (2) frequency of non-specific skin conductance responses (NS-SCR).

SECONDARY OUTCOMES:
Children's Dental Behavioral Rating Scale (CDBRS) | Videorecorded throughout dental cleaning (approximately 10-45 minutes); coded during first five minutes of dental prophylaxis.
  The Children's Dental Behavioral Rating Scale (CDBRS) evaluates overt distress behaviors exhibited by children in the dental office. The child's behavior is videotaped during the dental cleaning; the first five minutes of prophylaxis are coded from the video data at a later date. Coding included marking the presence or absence of three distress behaviors (mouth movement, head movement, forehead movement) and the presence or absence and the severity of two distress behaviors (whimper/cry/scream, verbal stall or delay) during each one-minute interval of the five minute video. Significant inter-rater reliability by two trained raters on a sample of children with and without ASD was obtained. The raw score (0-45) was converted, via Rasch analysis, to a scale score of 1-100.
Number of hands used to restrain child | Recorded throughout the dental cleaning (approximately 10-45 minutes)
  The number of hands required to restrain the child during the dental cleaning experience was also utilized as a measure of uncooperative behavior. This variable was recorded on researcher notes during the dental cleaning and was verified using the videotape of the dental cleaning. Scoring included presence/absence as well as the number of hands used for restraint purposes during the cleaning.
Frankl Scale | Completed at the end of each dental cleaning (approximately 10-45 minutes)
  The Frankl Scale was completed by the dentist following the dental cleaning. This one-item Likert Scale ranges from 1 (definitely negative) to 2 (negative) to 3 (positive) to 4 (definitely positive). This assessment has high inter-rater reliability and moderate validity and has been used to measure the behavior of children with ASD.
The Anxiety and Cooperation Scale (A & C Scale) | Completed at the end of each dental cleaning (approximately 10-45 minutes)
  The Anxiety and Cooperation Scale (A & C Scale) has been shown to assess children's anxiety, fear, and cooperation as rated by dentists, and has good established reliability and validity. Following a routine dental cleaning, the dentist rated overall patient behavior during treatment using a one-item Likert scale ranging from 0 (relaxed, smiling, demonstrates desired behavior, complies with demands) to 5 (out of control, loud crying, reverts to primitive flight responses, physical restraint required).
Time | Time from beginning to end of dental cleaning (approximately 10-45 minutes); recorded for each visit
  The length of time to complete the dental cleaning. Used for cost-analysis of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Cermak, EdD, Principal Investigator — University of Southern California

REFERENCES:
- [Derived] Chaspari T, Tsiartas A, Stein Duker LI, Cermak SA, Narayanan SS. EDA-gram: designing electrodermal activity fingerprints for visualization and feature extraction. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:403-406. doi: 10.1109/EMBC.2016.7590725. PMID 28268358
- [Derived] Cermak SA, Stein Duker LI, Williams ME, Dawson ME, Lane CJ, Polido JC. Sensory Adapted Dental Environments to Enhance Oral Care for Children with Autism Spectrum Disorders: A Randomized Controlled Pilot Study. J Autism Dev Disord. 2015 Sep;45(9):2876-88. doi: 10.1007/s10803-015-2450-5. PMID 25931290
- [Derived] Cermak SA, Stein Duker LI, Williams ME, Lane CJ, Dawson ME, Borreson AE, Polido JC. Feasibility of a sensory-adapted dental environment for children with autism. Am J Occup Ther. 2015 May-Jun;69(3):6903220020p1-10. doi: 10.5014/ajot.2015.013714. PMID 25871593
- [Derived] Chaspari T, Tsiartas A, Stein LI, Cermak SA, Narayanan SS. Sparse representation of electrodermal activity with knowledge-driven dictionaries. IEEE Trans Biomed Eng. 2015 Mar;62(3):960-71. doi: 10.1109/TBME.2014.2376960. Epub 2014 Dec 4. PMID 25494494
- [Derived] Stein LI, Lane CJ, Williams ME, Dawson ME, Polido JC, Cermak SA. Physiological and behavioral stress and anxiety in children with autism spectrum disorders during routine oral care. Biomed Res Int. 2014;2014:694876. doi: 10.1155/2014/694876. Epub 2014 Jul 10. PMID 25114916